CLINICAL TRIAL: NCT03362866
Title: Epidemiology of Hepatitis B, C and Delta in Reunion Island
Acronym: HEPEPID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/CHU/14
Record Dates: First submitted 2017-11-24; First posted 2017-12-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis B; Hepatitis C; Hepatitis D
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Viral hepatitis B, C and Δ represent a global public health problem for which France was very early mobilized. Despite this, in its foreword, the Dhumeaux report on "Management of people infected with hepatitis B or hepatitis C viruses" identifies a residual area of weakness in this care that is the incomplete regional epidemiological data in the Overseas Territories. The specific ethno-socio-cultural characteristics of these territories make it difficult to transpose data from the mainland France. This study aims at improving our knowledge on the characteristics of patients with hepatitis B, C and Δ in Reunion Island, their follow-up, their evolution and complications.

ELIGIBILITY:
Inclusion Criteria:

Major patient

* with confirmed HBsAg and / or anti HCV positive Ab
* residing in Reunion Island
* followed in one of the participating centers

Exclusion Criteria:

• Patient carrying isolated anti HBc antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatitis B, C, D patients in Reunion Island
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with hepatitis B, C and Δ in Reunion | Up to 5 years
  Hepatitis diagnosis will be made according to the ongoing guidelines in France (referred by the National AIDS and Hepatitis Research Agency (ANRS)

IPD SHARING:
Plan to Share IPD: No